CLINICAL TRIAL: NCT02751385
Title: A Phase I Trial to Investigate the Effect of Nintedanib on the Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Patients With Non-small Cell Lung Cancer
Brief Title: Investigation of the Effect of Nintedanib on the Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated- Study halted due to low recruitment.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1199.238; 2015-005664-41 (EudraCT Number)
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ethinyl estradiol, levonorgestrel drug combination; nintedanib

ARMS (1):
- All Patients (Experimental): Microgynon alone in Period 1 then with Nintedanib in Period 2
  Interventions: Drug: Microgynon; Drug: Nintedanib

INTERVENTIONS:
Drug: Microgynon
Drug: Nintedanib

SUMMARY:
Investigate the effect of multiple oral doses of nintedanib on the single dose kinetics of a combination of ethinylestradiol and levonorgestrel (Microgynon®)

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Female patients 18 years or older at screening
* Female patient is postmenopausal or surgically sterilised
* Patient with locally advanced, metastatic or locally recurrent non-small cell lung cancer with histology of adenocarcinoma
* Nintedanib (Vargatef®) is planned to be prescribed in accordance with the marketing authorisation (SmPC)
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial

Exclusion criteria:

* Any contraindication to nintedanib (Vargatef®), ethinylestradiol or levonorgestrel (Microgynon®), as specified in the respective labels
* Use of hormone containing contraceptives (including vaginal and intrauterine devices and including hormone replacement therapy) within 30 days prior to first administration of Microgynon®
* Systemic use of drugs known to induce (e.g. rifampicin, St. John's Wort, carbamazepine) or to inhibit (e.g. azole antimycotics, macrolides) CYP3A4 within 7 days prior to first trial drug administration until last pharmacokinetic(PK)-sampling in the trial. Exception: allowed is the intake of corticosteroids as docetaxel (pre)medication
* History of major thrombotic or clinically relevant major bleeding event in the past 6 months
* Persistence of clinically relevant therapy related toxicities (i.e. > Common Terminology Criteria for Adverse Events [CTCAE] grade 2) from previous chemotherapy and/or radiotherapy
* Treatment with other investigational drugs or treatment in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the trial drugs
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to first treatment within the trial and without complete wound healing
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patients unable to comply with the protocol
* Previous enrolment in this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Klinikum Chemnitz gGmbH, Chemnitz, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I study to investigate the effect of multiple oral doses of nintedanib on the single dose kinetics of a combination of ethinylestradiol and levonorgestrel (Microgynon®) in patients with non-small cell lung cancer.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all subjects met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Microgynon®: Patients were orally administered one tablet of Microgynon® (combination of 30 microgram ethinylestradiol and 150 microgram levonorgestrel per tablet) after a standardised breakfast in Period 1.
- Microgynon® With Nintedanib: Patients were orally administered one tablet of Microgynon® after continuous 2x2 nintedanib soft gelatine capsule containing 100 mg per day (with dose reduction to 2x1 capsule containing 150 mg, if required) for at least 7 consecutive days in Period 2.
  Nintedanib was to be taken continuously throughout Period 2. In case of a temporary interruption of nintedanib intake, patients could receive Microgynon® in Period 2 only if they had taken nintedanib for at least 7 consecutive days before intake of Microgynon®.
Period: Period 1
Arm/Group | Microgynon® | Microgynon® With Nintedanib
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Microgynon® | Microgynon® With Nintedanib
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS)- This patient set includes all patients in the Entered Set (ES) who were documented to have received one dose of study drug.
Groups:
- All Patients: Patients were orally administered one tablet of Microgynon® (combination of 30 microgram ethinylestradiol and 150 microgram levonorgestrel per tablet) after a standardised breakfast in Period 1.
  Patients were orally administered one tablet of Microgynon® after continuous 2x2 nintedanib soft gelatine capsule containing 100 mg per day (with dose reduction to 2x1 capsule containing 150 mg, if required) for at least 7 consecutive days in Period 2.
  Nintedanib was to be taken continuously throughout Period 2. In case of a temporary interruption of nintedanib intake, patients could receive Microgynon® in Period 2 only if they had taken nintedanib for at least 7 consecutive days before intake of Microgynon®. Same subjects were continued to Period 2, hence baseline characteristics are presented by Period 1.
Arm/Group | All Patients
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: TS
  years | 67.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 2
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 2
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 2
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the the Ethinylestradiol and Levonorgestrel in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC 0-tz) for ethinylestradiol and levonorgestrel after a single dose of the combination of ethinylestradiol and levonorgestrel. In Period 1, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h and 72h after drug administration of Microgynon®. Nintedanib in Period 2 was started at least 7 days before Microgynon® administration.
  In Period 2, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 11.55h, 23.55h, 47.55h and 71.55h after drug administration of Microgynon®.
Time Frame: Please refer to description section for the details about the actual sampling time points
Population: Pharmacokinetic Set (PKS): This analysis set includes all patients in the Treated Set (TS) who contributes only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/mililiter
Arm/Group | Microgynon® | Microgynon® With Nintedanib
Number analyzed (Participants) | 2 | 2
picogram*hour/mililiter
  Ethinylestradiol: number analyzed (Participants) | 2 | 1
  Ethinylestradiol | 410 (6.61) | 348 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.
  Levonorgestrel: number analyzed (Participants) | 2 | 1
  Levonorgestrel | 41500 (11.0) | 43600 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.

2. Primary Outcome: Maximum Measured Concentration (Cmax) of Ethinylestradiol and Levonorgestrel
Description: Maximum blood concentrations (Cmax) for ethinylestradiol and levonorgestrel after a single dose of the combination of ethinylestradiol and levonorgestrel. In Period 1, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h and 72h after drug administration of Microgynon®. Nintedanib in Period 2 was started at least 7 days before Microgynon® administration.
  In Period 2, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 11.55h, 23.55h, 47.55h and 71.55h after drug administration of Microgynon®.
Time Frame: Please refer to description section for the details about the actual sampling time points
Population: Pharmacokinetic Set (PKS): This analysis set includes all patients in the TS who contributes only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter[pg/mL]
Arm/Group | Microgynon® | Microgynon® With Nintedanib
Number analyzed (Participants) | 2 | 2
picogram/milliliter[pg/mL]
  Ethinylestradiol: number analyzed (Participants) | 2 | 1
  Ethinylestradiol | 32.6 (3.04) | 36.9 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.
  Levonorgestrel: number analyzed (Participants) | 2 | 1
  Levonorgestrel | 2680 (23.2) | 1630 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.

3. Secondary Outcome: Area Under the Concentration-time Curve of the Ethinylestradiol and Levonorgestrel in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity).
Description: Area under curve from zero to infinity (AUC0-∞) for ethinylestradiol and for levonorgestrel after intake of a single dose of the combination of ethinylestradiol and levonorgestrel. In Period 1, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 48h and 72h after drug administration of Microgynon®. Nintedanib in Period 2 was started at least 7 days before Microgynon® administration.
  In Period 2, blood samples were collected at pre-dose at 0.35 hour (h) and at 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 11.55h, 23.55h, 47.55h and 71.55h after drug administration of Microgynon®.
Time Frame: Please refer to description section for the details about the actual sampling time points
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Microgynon® | Microgynon® With Nintedanib
Number analyzed (Participants) | 2 | 1
pg*h/mL
  Ethinylestradiol | 503 (0.394) | 580 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.
  Levonorgestrel | 54500 (9.52) | 57600 (NA) — Only one patient was analysed, thus Geometric coefficient of variation (gCV) was not calculated.

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after the last drug administration. Up to 13 days for Microgynon. From first drug administration until 30 days after the last drug administration. Up to 34 days for nintedanib.
Groups:
- Loading Nintedanib: Patients on nintedanib loading phase
- Nintedanib+Microgynon®: Patients were orally administered one tablet of Microgynon® after continuous 2x2 nintedanib soft gelatine capsule containing 100 mg per day (with dose reduction to 2x1 capsule containing 150 mg if required) for at least 7 consecutive days in Period 2. Nintedanib was to be taken continuously throughout in Period 2. In case of a temporary interruption of nintedanib intake, patients could receive Microgynon® in Period 2 only if they have taken nintedanib for at least 7 consecutive days before intake of Microgynon®.
- Nintedanib: Patients administered with nintedanib
Arm/Group | Microgynon® | Loading Nintedanib | Nintedanib+Microgynon® | Nintedanib
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 1/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon® (N=2) | Loading Nintedanib (N=2) | Nintedanib+Microgynon® (N=2) | Nintedanib (N=2)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT02751385/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02751385/SAP_001.pdf